CLINICAL TRIAL: NCT03411980
Title: An Open-label, Single-dose Study to Evaluate the Pharmacokinetics and Safety of Vilaprisan in Subjects With Decreased Renal Function in Comparison With Matched Subjects With Normal Renal Function
Brief Title: Pharmacokinetics and Safety of Vilaprisan in Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 16524
Record Dates: First submitted 2018-01-22; First posted 2018-01-26 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-12

CONDITIONS: Uterine Fibroids; Endometriosis
Keywords: Pharmacokinetics
MeSH Terms: conditions — Leiomyoma; Endometriosis | interventions — vilaprisan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Subjects with moderately decreased renal function (Experimental): Subjects with moderate renal impairment with an estimated glomerular filtration rate (eGFR) of 30 to 59 mL/min/1.73 m*2 according to the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula.
  Interventions: Drug: Vilaprisan (BAY1002670)
- Subjects with severely decreased renal function (Experimental): Subjects with severe renal impairment not on dialysis with an eGFR <30 mL/min/1.73 m*2 (CKD-EPI formula).
  Interventions: Drug: Vilaprisan (BAY1002670)
- Control subjects with normal renal function (Experimental): Subjects with an eGFR ≥90 mL/min/1.73 m*2 (CKD-EPI formula) who are matched based on sex, age, race and weight.
  Interventions: Drug: Vilaprisan (BAY1002670)

INTERVENTIONS:
Drug: Vilaprisan (BAY1002670) — Single oral dose (1 x 2 mg immediate-release, film-coated tablet)

SUMMARY:
The purpose of the study is to evaluate the pharmacokinetics of vilaprisan in subjects with moderate to severe renal impairment compared with matched subjects with normal renal function.

DETAILED DESCRIPTION:
This is a multiple-center, open-label, non-randomized, single-dose study in 3 parallel groups of subjects with moderately or severely impaired renal function or normal renal function matched with regard to sex, age, race and weight. PK blood and urine sampling for determination of vilaprisan concentrations in plasma and urine, respectively, will be preformed at pre-defined time points up to 14 days post-dose. Safety and tolerability will be assessed through adverse events, clinical laboratory tests, vital signs, 12-lead electrocardiograms and physical examinations.

ELIGIBILITY:
Inclusion Criteria:

* BMI: 18 to 40 kg/m*2 (inclusive)
* Decreased renal function, as assessed at screening, based on serum creatinine and calculated according to the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula, either:

Moderately impaired renal function: eGFR: 30 to 59 mL/min/1.73 m*2; or Severely impaired renal function: eGFR <30 mL/min/1.73 m*2 but not on dialysis

- Normal renal function, as assessed at screening and based on serum creatinine according to the CKD-EPI formula: eGFR ≥90 mL/min/1.73 m*2

Exclusion Criteria:

* Any relevant disease within 4 weeks prior to study drug administration including infections and acute gastrointestinal diseases (vomiting, diarrhea, constipation) requiring medical treatment.
* Severe cerebrovascular or cardiac disorders less than 6 months prior to study drug administration, e.g. stroke, myocardial infarction, unstable angina pectoris, percutaneous transluminal coronary angioplasty or coronary artery bypass graft, congestive heart failure of Grade III or IV according to New York Heart Association, or arrhythmia requiring antiarrhythmic treatment.
* Malignancy diagnosed or treated within the past 5 years. This does not include adequately treated basal cell carcinoma or localized squamous cell carcinoma of the skin.
* Acute renal failure or acute nephritis within the past 2 years.
* Pregnancy or lactation.
* Use of CYP3A4 inducers from 2 weeks before study drug administration until last day of blood sampling for PK after study drug administration, including grapefruits.
* Insufficiently controlled diabetes mellitus with fasting blood glucose >220 mg/dL or HbA1c >10%.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2018-10-10 (Actual); Study Completion 2019-02-06 (Actual)

PRIMARY OUTCOMES:
Area under the concentration versus time curve from zero to infinity after single (first) dose (AUC) of BAY1002670 | -1hour (h), 30minutes (min), 1h, 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 12h ,16h, 1day (d), 2d, 3d, 4d, 7d, 10d, 14d
  Area under the concentration versus time curve from zero to the last data point above the lower limit of quantitation [AUC(0-tlast)], if AUC cannot be estimated in all subjects.
  In subjects with normal and moderately reduced renal function.
Maximum observed drug concentration in measured matrix after single dose administration (Cmax) of BAY1002670 | -1h, 30min, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 12h ,16h, 1d, 2d, 3d, 4d, 7d, 10d, 14d
  In subjects with normal and moderately reduced renal function.

SECONDARY OUTCOMES:
Number of participants with adverse events | Up to 6 weeks
  In subjects with normal, moderately, and severely reduced renal function.
AUC | -1h, 30min, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 12h ,16h, 1d, 2d, 3d, 4d, 7d, 10d, 14d
  In subjects with normal, moderately, and severely reduced renal function.
unbound AUC (AUCu) | -1h, 30min, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 12h ,16h, 1d, 2d, 3d, 4d, 7d, 10d, 14d
  In subjects with normal, moderately, and severely reduced renal function.
Cmax | -1h, 30min, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 12h ,16h, 1d, 2d, 3d, 4d, 7d, 10d, 14d
  In subjects with normal, moderately, and severely reduced renal function.
Unbound Cmax (Cmax,u) | -1h, 30min, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 12h ,16h, 1d, 2d, 3d, 4d, 7d, 10d, 14d
  In subjects with normal, moderately, and severely reduced renal function.
Apparent oral clearance (CL/F) | -1h, 30min, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 12h ,16h, 1d, 2d, 3d, 4d, 7d, 10d, 14d
  In subjects with normal, moderately, and severely reduced renal function.
Unbound CL/F (CLu/F) | -1h, 30min, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 12h ,16h, 1d, 2d, 3d, 4d, 7d, 10d, 14d
  In subjects with normal, moderately, and severely reduced renal function.
Half-life associated with the terminal slope (t1/2) | -1h, 30min, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 12h ,16h, 1d, 2d, 3d, 4d, 7d, 10d, 14d
  In subjects with normal, moderately, and severely reduced renal function.
Renal clearance (CLR) | -1h, 30min, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 12h ,16h, 1d, 2d, 3d, 4d, 7d, 10d, 14d
  In subjects with normal, moderately, and severely reduced renal function.
Fraction of free (unbound) drug in plasma (fu) | -1h, 30min, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 12h ,16h, 1d, 2d, 3d, 4d, 7d, 10d, 14d
  In subjects with normal, moderately, and severely reduced renal function.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Clinical Pharmacology of Miami, Inc., Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida

REFERENCES:
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/